CLINICAL TRIAL: NCT00002935
Title: A Phase II Study of the Safety and Efficacy of Photodynamic Therapy in Carcinoma in Situ of the Esophagus
Brief Title: Photodynamic Therapy in Treating Patients With Early Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS 93-23; RPCI-DS-93-23
Record Dates: First submitted 1999-11-01; First posted 2003-10-22 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Esophageal Cancer
Keywords: stage 0 esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: porfimer sodium

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. This may be an effective treatment for esophageal cancer.

PURPOSE: Phase II trial to study the effectiveness of photodynamic therapy in treating patients with Barrett's esophagus who have in situ esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of photodynamic therapy (PDT) using porfimer sodium (Photofrin) and controlled uniform laser light in patients with carcinoma in situ in Barrett's esophagus or severe dysplasia in Barrett's esophagus. II. Evaluate the safety of the treatment on this patient.

OUTLINE: This is a noncomparative study. PDT consists of IV porfimer sodium followed 40-50 hours later by laser red light delivered by optic fibers passed through the biopsy channel of an endoscope. Retreatment, if necessary, consists of up to 3 injections at least 30 days apart and up to 6 laser light treatments, with a maximum of 2 following each injection. Patients are followed monthly for 4 months, and then periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary, stage 0 carcinoma in situ (CIS) in conjunction with Barrett's esophagus or severe dysplasia in Barrett's esophagus who are medically unsuitable for or have refused surgery Previously biopsied Barrett's mucosa with areas of severe dysplasia and/or CIS

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky greater than 50% Life expectancy: Not specified Hematopoietic: WBC at least 2,000/mm3 Platelet count at least 50,000/mm3 Hepatic: No porphyria or hypersensitivity to porphyrins Bilirubin no greater than 3.0 mg/dL Alkaline phosphatase no greater than 3 times ULN SGOT no greater than 3 times ULN PT no greater than 1.5 times the upper limit of normal (ULN) Renal: Creatinine no greater than 3.0 mg/dL Other: No contraindication to endoscopy Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent chemotherapy At least 1 month since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiation therapy No concurrent laser therapy At least 1 month since prior radiation therapy At least 1 month since prior laser therapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1995-10; Primary Completion 2006-08 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector R. Nava, MD, FACS, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States